CLINICAL TRIAL: NCT06874543
Title: The Effect of Visceral Osteopathic Manual Therapy Methods in Women With Stress Urinary Incontinence
Brief Title: Visceral Osteopathic Manual Therapy Methods in Women With Stress Urinary Incontinence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Rumeli University (Other)
Responsible Party: Principal Investigator, NEZAHAT AKIN, Principal investıgator physiotherapist, Istanbul Rumeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRU-FTR-NA-01
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Osteopathic Manipulative Treatment (OMT)
Keywords: Urinary Stress Incontinence; Osteopathic Manipulative Treatment (OMT); Quality of Life
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: 40 volunteer female patients who applied to the polyclinics with complaints of urinary incontinence, diagnosed with SUI by specialist doctors, aged between 18 and 70, who can communicate in Turkish, who can read and write, and who can accept verbal warnings will be included. Patients with prolapse, vaginal and urinary system infection or malignancy, neurological damage, or who have had a disease or surgery that may cause incontinence, and pregnant women will be excluded from the study. Patients will be randomly divided into 2 groups as treatment and control, with 20 people in each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Study group visceral osteopathic manual therapy method will be applied (Active Comparator): In the study, relaxation techniques, hepato-gastric ligamentum mobilization, pyloric valve mobilization, sphincter odi mobilization, sphincter ilio-jejunum mobilization, cecal valve mobilization, iliopsoas and iliacus mobilization, peritoneal mobilization, intestine, kidney, bladder, stomach, liver and bladder organ mobilizations will be applied to the experimental group patients as VOMT program. Until the next session, bladder mobilization will be taught as a home program and they will be asked to do it every day. After VOMT is applied by the physiotherapist once a week, a total of 4 times, the evaluation scales will be applied again. In order to see the long-term effect, the patients will be evaluated again in the first month and the third month after the end of the treatment. The forms will be filed as pre-treatment, post-treatment, first month and third month data and will be entered into the computer and recorded.
  Interventions: Other: visceral osteopathic manual therapy
- Group 2: Evaluation scales will be applied to control group patients on the first day, and the scale (No Intervention): They were evaluated on the first application day and followed up ten times in parallel with the study group, at 1 month, 2 months and 4 months, a total of 4 times.

INTERVENTIONS:
Other: visceral osteopathic manual therapy — In the study, relaxation techniques, hepato-gastric ligamentum mobilization, pyloric valve mobilization, sphincter odi mobilization, sphincter ilio-jejunum mobilization, cecal valve mobilization, iliopsoas and iliacus mobilization, peritoneal mobilization, intestine, kidney, bladder, stomach, liver and bladder organ mobilizations will be applied to the experimental group patients as VOMT program. Until the next session, bladder mobilization will be taught as a home program and they will be asked to do it every day. After VOMT is applied by the physiotherapist once a week, a total of 4 times, the evaluation scales will be applied again. In order to see the long-term effect, the patients will be evaluated again in the first month and the third month after the end of the treatment. The forms will be filed as pre-treatment, post-treatment, first month and third month data and will be entered into the computer and recorded
  Arms: Group 1: Study group visceral osteopathic manual therapy method will be applied

SUMMARY:
The aim of this study is to evaluate the effect of visceral osteopathic manual therapy method for stress urinary incontinence in female patients. As a result of the study, the effect of visceral osteopathic manual therapy fascial release on bladder control, quality of life and flexibility will be evaluated.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is an important health problem that occurs when continence cannot be achieved and negatively affects the lives of individuals according to the International Continence Society (ICS). Stress urinary incontinence (SUI), one of the most common types of UI, is a problem that occurs during coughing, laughing, sneezing, exercise (one of which is caused by increased intra-abdominal pressure (Valsalva maneuver) and shows a steady increase in women with age. The aim in the treatment of SUI is to ensure that patients regain their continence skills. In recent years, conservative treatment methods have been preferred more in the treatment of SUI due to their ease of application and low cost. It is thought that Osteopathic Manual Therapy (OMT) reduces the negative effects of musculoskeletal pain and dysfunction on body systems, improves respiratory mechanics, venous and lymphatic drainage, and accordingly supports homeostasis and optimizes functions.

In this study, it is planned to investigate the effect of the visceral system and visceral fascia on SUI.

It is thought that the fascia surrounding the internal organs can be loosened and systematic diseases can be affected with the visceral osteopathic manual therapy (VOMT) method, which is among the osteopathic manual therapy methods.

Within the scope of the study, 40 volunteer female patients diagnosed with SUI will be evaluated and randomly divided into 2 groups. Day 1 evaluation scales will be applied to both groups, VOMT methods will be applied to the experimental group a total of four times a week, and bladder mobilization will be given as a home program, and no application will be made to the control group. Both groups will be re-evaluated in months 1 and 4. The inadequacy of studies conducted on this subject was an important factor in choosing this method.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between the ages of 18 and 70
* Being able to communicate in Turkish
* Being able to read and write
* Being able to understand and follow verbal prompts
* Being willing to participate in the study

Exclusion Criteria:

* Pregnancy
* Presence of prolapse
* Presence of vaginal and urinary system infection or malignancy
* Presence of neurological damage
* Having had any disease that may cause incontinence
* Having had surgery for SUI or urogynecological reasons in the last 2 months.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — • Being a woman between the ages of 18 and 70
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
pad test | 4 months after registration
  In this test, standardized by the International Incontinence Society, the patient is asked to place a clean pad in their underwear and then do some activities in order. These activities are done in the following order;
  * Drink 500 ml of water,
  * Walk for 30 minutes,
  * Sit down and stand up 10 times in the 45th minute, cough 10 times,
  * Run for 1 minute, then pick up objects from the ground without resting,
  * Finally, wash your hands for 3 minutes. After the pad is placed, the pad is taken out in the 60th minute and weighed on a precision scale in grams (gr), the dry weight is subtracted from the wet weight and the difference is recorded as data.
feeling of dryness (VAS) | 4 months after registration
  The effect of UI on the woman's life and the feeling of dryness she perceived were assessed with VAS. In the VAS assessment, the woman was asked to mark the intensity of her feeling on a 10 cm line. While the left side of the line meant "it has no effect on my life" or "I feel dry", it was stated that this "intensity increases" towards the right of the line and the far right side meant "it affects my life a lot" or "I feel constantly wet". The marked point was measured with a ruler and recorded in cm.
"International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) | 4 months after registration
  In order to ensure standardization in pre- and post-treatment evaluations in clinical studies, there is a need for standardized questionnaire forms regarding urinary incontinence. These forms should be short, understandable and purposeful. Among the questionnaire forms regarding urinary incontinence, the "International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) is thought to meet all these requirements in this regard.
Incontinence Quality of Life Questionnaire (I-QOL): | 4 months after registration
  According to this survey, individuals are asked 28 questions about their daily lives and psychosocial situations. Individuals are asked to answer each question as no (0), mild (1), moderate (2) and severe (3). The score obtained from the twenty-eight questions is recorded as a total score. A high score means that the quality of life is negatively affected.

SECONDARY OUTCOMES:
Incontinence severity level | 4 months after registration
  In order to determine the severity of incontinence, the incontinence severity level is determined as mild, moderate and severe according to the frequency of urine leakage (Pages I-H, Jahr S & al.lari, 2001);
  * Mild incontinence (grade 1): Incontinence that occurs involuntarily during laughing, coughing, sneezing or heavy exercise
  * Moderate incontinence (grade 2): Incontinence that occurs involuntarily during light activities, walking or carrying objects
  * Severe incontinence (grade 3): Incontinence that occurs even when standing up but not at rest
Flexibility tests(trunk extension flexibility) | 4 months after registration
  In individuals experiencing incontinence, the flexibility of the abdominal region, back region and lower extremity should be evaluated. To evaluate trunk flexibility, trunk extension flexibility, trunk lateral flexion flexibility tests, and the Sit and Reach Test can be used to evaluate lower extremity and trunk flexibility.
Body temperature | 4 months after registration
  Body temperature should be measured with an infrared thermometer 5 cm above and below the umbilicus and the values should be recorded.
Flexibility tests( trunk lateral flexion flexibility) | 4 months after registration
  In individuals experiencing incontinence, the flexibility of the abdominal region, back region and lower extremity should be evaluated. To evaluate trunk flexibility, trunk extension flexibility, trunk lateral flexion flexibility tests, and the Sit and Reach Test can be used to evaluate lower extremity and trunk flexibility.
Flexibility tests( Sit and Reach Tes) | 4 months after registration
  In individuals experiencing incontinence, the flexibility of the abdominal region, back region and lower extremity should be evaluated. To evaluate trunk flexibility, trunk extension flexibility, trunk lateral flexion flexibility tests, and the Sit and Reach Test can be used to evaluate lower extremity and trunk flexibility.

OTHER OUTCOMES:
Demographic data form | 4 months after registration
  A detailed history and a complete physical examination are the first and most important steps used in the evaluation of the patient. Personal information such as age, weight, occupation, and educational status should be questioned with the demographic data form, where information about the person can be questioned. The signs and symptoms of UI, and the presence of urinary incontinence that occurs after an increase in intra-abdominal pressure such as coughing, sneezing, or laughing should be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: ALİ CIMBIZ, PROFESSOR, Study Director — Istanbul Rumeli University
Locations (1):
- Istanbul Rumeli University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No